CLINICAL TRIAL: NCT05167123
Title: Radiographic and Clinical Evaluation of Indirect and Direct Pulp Capping in Primary Molars Using TheraCal (LC)
Brief Title: Pulp Capping in Primary Molars Using TheraCal (LC)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yomna Hussein Moselhy, Principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-RECIM041919
Record Dates: First submitted 2021-09-28; First posted 2021-12-22 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Deep Caries; Indirect Pulp Capping; Direct Pulp Capping; Reversible Pulpitis; Decayed Teeth; Vital Pulp Therapy
Keywords: IPC , DPC
MeSH Terms: conditions — Dental Caries | interventions — TheraCal

STUDY DESIGN:
Intervention Model Description: Simple parallel randomization was performed by using computerized random numbers
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and the outcome assessor were blinded. The primary investigator blinding was impossible
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indirect Pulp Capping (Experimental): TheraCal (LC) will be applied to affected dentin after excavation of infected dentin
  Interventions: Drug: Light cured tri-calcium silicate base material
- Direct Pulp Capping (Experimental): TheraCal (LC) will be applied to pinpoint pulp exposures (less than 1mm ) in vital pulps surrounded by sound dentin.
  Interventions: Drug: Light cured tri-calcium silicate base material

INTERVENTIONS:
Drug: Light cured tri-calcium silicate base material — TheraCal (LC) (BISCO Inc., Schamburg, IL, USA) was introduced in (2011), are available commercially as flowable cement applicable via syringe
  Other Names: TheraCal (LC)

SUMMARY:
A randomized clinical trial that aims to evaluate clinical and radiographic success rates of indirect pulp capping and direct pulp capping in primary molars with reversible pulpitis using a light-cured tri-calcium silicate base material (TheraCal (LC)).

DETAILED DESCRIPTION:
Participating primary molars will be randomly allocated to one of the following groups: Indirect pulp capping group or Direct pulp capping group. A light-cured tri-calcium silicate base material (TheraCal (LC) ) will be used in the two groups as a dressing material. Patients will be recruited from the outpatient clinic of the pediatric dentistry department, Faculty of Dentistry Ain Shams University. The participant will be recalled for follow-up assessments at 3, 6,9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 4-7 years.
2. Free medical history.
3. Complete physical and mental health.
4. Patient cooperation
5. restorable mandibular primary molars

Exclusion Criteria:

1. Clinical symptoms or irreversible pulpitis as (spontaneous pain, throbbing pain)
2. Soft tissue swelling, draining fistula or sinus tracts.
3. Tenderness to percussion.
4. Pathological Tooth mobility.
5. Widening of periodontal membrane space

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
recording signs and symptoms through clinical examination | one year follow-up
  All the primary molars participating in this study will be examined clinically under the illumination of dental unit, percussion and palpation test will be performed to ensure absence of any sign and symptoms of irreversible pulpitis or nectrotic pulp during follow -up period.

SECONDARY OUTCOMES:
recording pathological Changes in Radiographic examination | one year follow-up
  All the primary molars participating in this study will be examined radiographically every (3,6,9,12 months) to ensure the absence of any pathological changes .
Evaluation of TheraCal (LC) as a pulp capping material | one year follow-up
  Clinical and radiographic examination will be done to each tooth participating in this study to evaluate the efficiency of TheraCal (LC) when used as a pulp capping material in primary molars .

CONTACTS AND LOCATIONS:
Overall Officials: Yomna Hussein Moselhy, M.Sc., Principal Investigator — Ain Shams University
Locations (3):
- Egypt (3):
  - Ain Shams University Faculy of Dentistry, Cairo
  - Department of pediatric dentistry - Ain Shams University, Cairo
  - Outpatient Clinic of the Department of Pediatric Dentistry, Ain Shams University, Cairo

IPD SHARING:
Plan to Share IPD: No